CLINICAL TRIAL: NCT05059756
Title: Percutaneous Tibial Nerve Stimulation and Pelvic Floor Rehabilitation in the Treatment of Childhood Constipation
Brief Title: PTNS and PFR in the Treatment of Childhood Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Shucheng Zhang, Professor, Shengjing Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A333
Record Dates: First submitted 2021-09-06; First posted 2021-09-28 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Constipation; Childhood ALL; Pelvic Floor Disorders
MeSH Terms: conditions — Constipation; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Pelvic Floor Disorders

STUDY DESIGN:
Intervention Model Description: Treatment group: PTNS and PFR treatment; Control group: ( Sham stimulation and PFR training)
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): PTNS and PFR (twice daily)
  Interventions: Device: PTNS
- Control group (Experimental): Sham PTNS and PFR (twice daily)
  Interventions: Device: Sham PTNS

INTERVENTIONS:
Device: PTNS — PTNS and PFR
  Other Names: PFR
  Arms: Treatment group
Device: Sham PTNS — Sham PTNS and PFR
  Other Names: PFR
  Arms: Control group

SUMMARY:
Constipation is the most common complaint in childhood, affecting an estimated 20% of children globally. At present, the treatment of children's constipation is full of challenges, and treatment methods are diverse.

Studies have shown that pelvic floor dysfunction is a common cause of intractable constipation in children. Zhang et al. have confirmed the role of pelvic floor dysfunction in pediatric constipation. At present, the main methods for pelvic floor dysfunction include surface electromyography and anorectal manometry which have been widely used in children with constipation and they are helpful for the diagnosis of pelvic floor dysfunction in children with constipation.

Sacral nerve electrical stimulation combined with pelvic floor rehabilitation is an effective method for the treatment of pelvic floor dysfunction. It offers a novel approach for the treatment of intractable constipation with pelvic floor dysfunction . At present, there are many methods for sacral nerve regulation. Percutaneous tibial nerve stimulation (PTNS), another peripheral nerve electrical stimulation approved by the United States Food and Drug Administration, has the same effect as sacral nerve regulation, and has the advantages of small trauma, safety, and convenience. However, there is still a lack of evidence-based support for the treatment of childhood constipation by PTNS combine with PFR. Therefore, in this study, a randomized, controlled, double-blind clinical trial was designed to confirm the efficacy and safety of PTNS combine with PFR in the treatment of childhood constipation.

DETAILED DESCRIPTION:
Constipation is the most common complaint in childhood, affecting an estimated 20% of children globally. At present, the treatment of childhood constipation is full of challenges, and treatment methods are diverse. For example, diet control, behavioral intervention and oral Laxative, bowl management, surgical treatment and other methods can be used for the treatment of childhood constipation. Therefore, a number of guidelines for constipation in children have been developed to regulate the treatment of constipation in children. Fiber intake and polyethylene glycol are recommended as the first line choice for constipation in North American and European guidelines. However, through clinical tests, the effectiveness of PEG3350 laxative and fiber does not last, or it does not work after long-term use. Therefore, additional treatment interventions are necessary. Zhang et al. applied traditional Chinese medicine to treat childhood constipation, which greatly improved the efficacy and reduced the recurrence rate, but there were still nearly 30% intractable constipation left, and other treatment methods were needed.

Studies have shown that secondary pelvic floor dysfunction is a common cause of intractable constipation in children. The incidence of pelvic floor dysfunction is high in children with constipation, and it has a great impact on the symptoms of constipation. Zhang et al. applied defecography to examine 76 children with constipation and found that there existed different pelvic floor dysfunction such as rectocele, puborectal muscle spasm, pelvic floor spasm syndrome and sigmoid hernia in the defecation of children with constipation. In addition, the pelvic floor dysfunction in children was mainly spastic, while in adults it was mainly flaccid. Although these results confirm the role of pelvic floor dysfunction in pediatric constipation, the pelvic floor function was not evaluated. At present, the main methods for pelvic floor function include surface electromyography and anorectal manometry.

Based on the above theory, Claire Zar-Kessler et al. completed a retrospective study of 69 children in which researchers compared the clinical outcome of patients who underwent pelvic floor physical therapy (n = 49) to control patients (n = 20) whom received only medical treatment (laxatives/stool softeners), determined by anorectal manometry and balloon expulsion testing and come to the conclusion that the new field of pelvic floor physical therapy is a safe and effective intervention for children with dyssynergic defecation causing or contributing to chronic constipation. In recent years, more and more studies have confirmed that childhood constipation is resulted from pelvic floor function.Also, it has been demonstrated that, after physical therapy, pelvic floor muscle was strengthened and it became fully continent of bowel in home and community settings. Therefore, constipation is one of the manifestations of pelvic floor dysfunction in children, surface electromyography assessment and anorectal manometry are helpful for the diagnosis of pelvic floor dysfunction in children.

Sacral nerve electrical stimulation combined with pelvic floor rehabilitation(PFR) is an effective method for the treatment of pelvic floor dysfunction. At present, there are many methods for sacral neuromodulation(SNM). Percutaneous sacral nerve stimulation is a effective method for sacral neuromodulation discovered in recent years. Studies have shown the efficacy of simultaneous SNM and PFR for the treatment of childhood constipation. This method is not only better than pelvic floor training and conventional treatment, but also safe and non-invasive. At present, there are many methods for SNM. Percutaneous tibial nerve stimulation (PTNS), another peripheral nerve electrical stimulation approved by the United States Food and Drug Administration, has the same effect as SNM, and has the advantages of small trauma, safety, and convenience. PTNS has become a very effective method for SNM in recent years. Carlo Vecchioli Scaldazza et al. demonstrates the effectiveness of PTNS in women with over active bladder, improving their pelvic floor function. The result suggests that percutaneous artificial stimulation combined with PFR can be used for the treatment of constipation, especially in those with secondary pelvic floor dysfunction.

Therefore, for the treatment of intractable constipation in children, it is also necessary to determine whether there is pelvic floor dysfunction involved. In the children with pelvic floor dysfunction, relieving the pelvic floor dysfunction is an important treatment principle for the treatment of constipation. PTNS in combination with PFR offers a novel approach for the treatment of pelvic floor dysfunction and intractable constipation. However, there is still a lack of evidence-based support for the treatment of childhood constipation by PTNS combine with PFR. In this study, a randomized, controlled, double-blind clinical trial was designed to confirm the efficacy and safety of PTNS combine with PFR in the treatment of childhood constipation.

ELIGIBILITY:
Inclusion Criteria:

* 4-14 years old;
* Meeting the Roman IV criteria for childhood constipation;
* After one course of PEG and one course of Chinese medicine treatment, it was ineffective;
* Pelvic floor surface electromyography (EMG) and 3-D manometry of the anus revealed pelvic floor dysfunction

Exclusion Criteria:meet one of the following criteria to be excluded:

* The onset of intestinal stenosis due to organic diseases (such as anal fissure, inflammation, intestinal polyps, intestinal adhesion, Crohn's disease, intestinal tuberculosis, tumor, etc.);
* constipation due to congenital diseases (such as congenital megacolon, sigmoid colon, etc.);
* Caused by metabolic endocrine diseases, neurological diseases and mental diseases;
* Those caused by systemic organic diseases;
* Patients diagnosed as outlet obstructive constipation and mixed functional constipation;
* Children with severe systemic diseases;
* Children with positive occult blood in stool routine examination;
* Children who refused to participate in PTNS combined with PFR.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2019-05-08 (Actual); Primary Completion 2021-12-08 (Actual); Study Completion 2021-12-08 (Actual)

PRIMARY OUTCOMES:
change of CSBMs (sub/week) from baseline | Baseline
  Rate of defecation without drugs or other auxiliary methods
change of CSBMs (sub/week) from baseline | at the end of 4-weeks PTNS and PFR treatment
  Rate of defecation without drugs or other auxiliary methods
change of CSBMs (sub/week) from baseline | at the end of 12 weeks follow-up
  Rate of defecation without drugs or other auxiliary methods
Satisfaction with bowel function | Baseline
  Satisfaction with bowel function was collected from the parents and defined as the number of which were satisfied with bowel function after the treatment (yes or no).
Satisfaction with bowel function Satisfaction with bowel function was collected from the parents and defined as whether they were satisfied with bowel function after the treatment (yes or no). | at the end of 4-weeks PTNS and PFR treatment
  Satisfaction with bowel function was collected from the parents and defined as the number of which were satisfied with bowel function after the treatment (yes or no).
Satisfaction with bowel function Satisfaction with bowel function was collected from the parents and defined as the number of which were satisfied with bowel function after the treatment (yes or no). | at the end of 12 weeks follow-up
  Satisfaction with bowel function was collected from the parents and defined as the number of which were satisfied with bowel function after the treatment (yes or no).

SECONDARY OUTCOMES:
Bowel movements the frequency of bowel movements per week | Baseline
  Rate of bowel movements per week;Incidence of constipation.
Bowel movements | at the end of 4-weeks PTNS and PFR treatment
  Rate of bowel movements per week;Incidence of constipation.
Bowel movements | at the end of 12 weeks follow-up
  Rate of bowel movements per week;Incidence of constipation.
Painful or hard bowel movements | Baseline
  The feelings of children during defecation;Rate of painful or hard bowel movements.
Painful or hard bowel movements | at the end of 4-weeks PTNS and PFR treatment
  The feelings of children during defecation;Rate of painful or hard bowel movements.
Painful or hard bowel movements | at the end of 12 weeks follow-up
  The feelings of children during defecation;Rate of painful or hard bowel movements.
Large diameter or scybalous stools | Baseline
  Appearance and wetness of stool; Rate of patients with large diameter or scybalous stools.
Large diameter or scybalous stools | at the end of 4-weeks PTNS and PFR treatment
  Appearance and wetness of stool; Rate of patients with large diameter or scybalous stools.
Large diameter or scybalous stools | at the end of 12 weeks follow-up
  Appearance and wetness of stool; Rate of patients with large diameter or scybalous stools.
Excessive volitional stool retention | Baseline
  Rate of children who intentionally control or reduce the frequency of defecation.
Excessive volitional stool retention | at the end of 4-weeks PTNS and PFR treatment
  Rate of children who intentionally control or reduce the frequency of defecation.
Excessive volitional stool retention | at the end of 12 weeks follow-up
  Rate of children who intentionally control or reduce the frequency of defecation.
Encopresis | Baseline
  Incidence of fecal incontinence
Encopresis | at the end of 4-weeks PTNS and PFR treatment
  Incidence of fecal incontinence
Encopresis | at the end of 12 weeks follow-up
  Incidence of fecal incontinence

CONTACTS AND LOCATIONS:
Overall Officials: Shucheng ZHANG, Study Chair — Shengjing Hospital; ZhengTong YU, Study Director — Shengjing Hospital
Locations (1):
- Shengjing Hospital, Shenyang, Liaoning, China

REFERENCES:
- [Background] Zar-Kessler C, Kuo B, Cole E, Benedix A, Belkind-Gerson J. Benefit of Pelvic Floor Physical Therapy in Pediatric Patients with Dyssynergic Defecation Constipation. Dig Dis. 2019;37(6):478-485. doi: 10.1159/000500121. Epub 2019 May 16. PMID 31096249
- [Result] Scaldazza CV, Morosetti C, Giampieretti R, Lorenzetti R, Baroni M. Percutaneous tibial nerve stimulation versus electrical stimulation with pelvic floor muscle training for overactive bladder syndrome in women: results of a randomized controlled study. Int Braz J Urol. 2017 Jan-Feb;43(1):121-126. doi: 10.1590/S1677-5538.IBJU.2015.0719. PMID 28124534